CLINICAL TRIAL: NCT05939479
Title: Impact of Antistaphylococcal Penicillins and Cefazolin on the Emergence of Resistance in French Hospitals
Brief Title: Antistaphylococcal Betalactam and Emergence of Resistance
Acronym: CePasR
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, LEFEVRE Benjamin, Doctor in the field of infectious diseases (MD PhD), Central Hospital, Nancy, France
Other Study IDs: 2023PI051
Record Dates: First submitted 2023-06-23; First posted 2023-07-11 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Bacterial Resistance; Methicillin-Sensitive Staphylococcus Aureus Infection
Keywords: cefazolin; antistaphylococcal penicillins; Methicillin-Sensitive Staphylococcus Aureus Infection; Bacterial Resistance

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Antistaphylococcal penicillins are recommanded as first-line agent in methicillin-suceptible Staphylococcus aureus bacteraemia. Several studies in progress are investigating the efficacy and safety of cefazolin compared with antistaphylococcal penicillins. Cefazolin has broader spectrum than antistaphylococcal penicillins. The hypothesis of this project is that cefazoline could be responsible for a higher rate of bacterial resistance. The aim is to study the association between the emergence of bacterial resistance and the consumption of cefazolin and antistaphylococcal penicillins.

ELIGIBILITY:
Inclusion Criteria: French hospitals which have collected their consumption and resistance data on the French national database named CONSORES (From 2019 to 2022)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients hospitalized in included French hospitals
Sampling Method: Non-Probability Sample
Enrollment: 644 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Association between the cefazolin/antistaphylococcal penicillins consumptions and the resistant bacteria emergence | Between the first january 2018 and the 31st december 2022
  The total consumption of antibiotics (expressed as number of Defined Daily Doses (DDD) per 1000 inhabitants per day) will be correlate with the resistant bacteria emergence (only incidence for each bacterial strain)

SECONDARY OUTCOMES:
Factors associated with the emergence of resistant bacteria | Between the first january 2018 and the 31st december 2022
  Factors associated with the emergence of resistant bacteria will be described by a Cox model: hospital size (number of beds), location in France, activities (intensive care, surgery, etc.), type of antibiotics and intensity of consumption expressed in number of defined daily doses (DDD).
Factors associated with the consumption of antibiotics | Between the first january 2018 and the 31st december 2022
  Factors associated with the emergence of resistant bacteria will be described by a Cox model: hospital size (number of beds), location in France, activities (intensive care, surgery, etc.) and type of bacterial strain indentified (resistant or not).
Evolution of resistance in French hospitals | Between the first january 2018 and the 31st december 2022
  For each year, bacterial resistance will be described, in France and in each hospital, in the form of a quantitative variable: number of resistant bacterial strains isolated for each year (number of resistant strains / total number of strains).
Evolution of antibiotics consumption in French hospitals | Between the first january 2018 and the 31st december 2022
  For each year, antibiotic consumption will be described, in France and in each hospital, in the form of a quantitative variable (expressed as number of Defined Daily Doses (DDD) per 1000 inhabitants per day)

CONTACTS AND LOCATIONS:
Locations (1):
- Lefevre, Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: No